

### **Informed Consent**

# INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH WITH OPTIONAL PROCEDURES

Phase II trial of sitravatinib plus nivolumab in patients with metastatic clear cell renal cell carcinoma who progress on prior treatment Acronym: SNAPI (Sitravatinib and Nivolumab After Prior Immunotherapy) 2021-0057

| Study Chair: Pavlos Msaoue | yl |
|----------------------------|-----------------------|
| Participant's Name | Medical Record Number |

This is an informed consent and authorization form for a research study. It includes a summary about the study. A more detailed description of procedures and risks is provided after the summary.

This research has been reviewed and approved by an Institutional Review Board (IRB - a committee that reviews research studies).

#### STUDY SUMMARY

The goal of this clinical research study is to learn if giving sitravatinib plus nivolumab can help control advanced kidney cancer after the disease has gotten worse (progressed) after receiving certain types of therapy. The safety of this drug combination will also be studied.

**This is an investigational study.** Sitravatinib is not FDA approved or commercially available. It is currently being used for research purposes only. Nivolumab is FDA approved and commercially available for the treatment of many types of cancer, including kidney cancer.

The study doctor can explain how the study drugs are designed to work.

The study drugs may help to control the disease. Future patients may benefit from what is learned. There may be no benefits for you in this study.

Your participation is completely voluntary. Before choosing to take part in this study, you should discuss with the study team any concerns you may have, including side effects (such as skin rash, fatigue, headache, high blood pressure, and/or diarrhea), potential expenses, and time commitment.

You can read a list of potential side effects below in the Possible Risks section of this consent.

You may continue to receive the study drugs for as long as the study doctor thinks it is in your best interest.

Sitravatinib and nivolumab will be provided at no cost to you while you are on study.

You may choose not to take part in this study. Instead of taking part in this study, you may choose to receive other investigational therapy, if available. The study doctor will discuss with you the possible risks and benefits of these treatments. You may choose not to have treatment for cancer at all. In all cases, you will receive appropriate medical care, including treatment for pain and other symptoms of cancer.

### 1. STUDY DETAILS

### **Screening Tests**

Signing this consent form does not mean that you will be able to take part in this study. You will have the below screening tests to help the doctor decide if you are eligible.

Within **6 months (180 days)** before your first dose of study drug, you will have an echocardiogram (ECHO) to check your heart function. If you have already had these tests performed as part of your standard care during this time, the results of that ECHO will be collected instead.

Within **28 days** before your first dose of study drugs:

- You will have a physical exam.
- You will have an MRI and/or CT scan of the chest, abdomen, and pelvis to check the status of the disease. You will have a CT scan or MRI of the brain. If the doctor thinks it is needed, you may also have an x-ray or bone scan.
- You will have an EKG to check your heart function.

Within **14 days** before your first dose of study drugs:

- You will have a physical exam.
- Blood (about 5 teaspoons) will be drawn for routine tests, which will include checking your blood sugar levels. You will fast (have nothing to eat or drink except water) for at least 8 hours before this blood draw.
- Urine will be collected for routine tests.
- You will complete 6 quality-of-life questionnaires. It should take about 1 hour to complete these questionnaires.
- If you can become pregnant, blood (about 2 teaspoons) or urine will be collected for a pregnancy test. To take part in this study, you must not be pregnant.

The study doctor will discuss the screening test results with you. If the screening tests show that you are not eligible to take part in the study, you will not be enrolled. Other options will be discussed with you.

Up to 88 participants will be enrolled in this multicenter study. Up to 40 will take part in MD Anderson.

### Study Drug Administration

Each study cycle is 28 days (4 weeks).

You will take **sitravatinib** capsules by mouth 1 time every day with a cup (about 8 ounces) of water. Each dose should be taken in the morning at about the same time each day. You should take sitravatinib at least 2 hours after and 1 hour before your next meal. For example, you can take your dose in the morning at least 1 hour before breakfast.

The capsules must be swallowed whole. Do not be chew, crush, or open them. If you vomit a dose of sitravatinib, do not take a "make up" dose. Wait and take your next dose as scheduled

You will be given a study drug diary to keep track of when you take each dose and if you miss or vomit any doses. You should return any empty study drug bottles or leftover study drug and the study drug diary to the clinic at the beginning of each cycle.

You will also receive **nivolumab** by vein over 30 minutes on Day 1 of each cycle.

You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

#### Study Visits

You may be able to have some of the below blood draws, urine collections, and physical exams done at a local doctor's office if that is more convenient for you. You will need to return to MD Anderson 1 time every cycle so the study doctor/study staff can check on you. This will be discussed with you.

### Day 1 of treatment (only Cycle 1):

• You will have an EKG to check your heart function 30-60 minutes before your first dose of sitravatinib. You will have a second EKG 5-9 hours after the dose.

# Day 15 of treatment (+/- 3 days, only Cycle 1):

You will have an EKG to check your heart function.

# **Every 4 weeks:**

- You will have a physical exam.
- Blood (about 1 teaspoon) will be drawn for routine tests, including tests to check certain hormone levels and the amount of fat in the blood. Tests of your hormone levels and fat levels will be done every 8 weeks for the first year then every 12 weeks after that.
- Urine will be collected for routine tests.
- At Week 8, 16, and 24, you will complete the same quality-of-life questionnaires that you completed at screening.

### Every 8 weeks for 1 year and then every 12 weeks after that:

• You will have an MRI and/or CT scan of the chest, abdomen, and pelvis to check the status of the disease. If the doctor thinks it is needed, you may also have an x-ray or bone scan.

**At Week 12 and then every 6 months after that**, you will have an ECHO. You may have this test more often if the doctor thinks it is needed.

If the disease gets worse, blood will be drawn for correlative research studies.

### **End-of-Treatment Visit**

About 30 days after your last dose of study drugs:

- You will have a physical exam.
- If the doctor thinks it is needed, you may have a CT or MRI scan of the chest, abdomen, and pelvis.

### Long-Term Follow-Up

You will be called by a member of the study staff every 3 months to ask how you are doing and if you have started any new anti-cancer treatments. This information may be collected from your medical record instead. This phone call should take about 5-10 minutes.

These calls will stop if you decide you no longer want to take part in this study.

# Other Testing

The study staff may ask you to take part in other MD Anderson research study (PA13-0291, PA17-0577, LAB02-152) for additional testing. The study doctor will discuss this with you and, if you decide to take part, you will sign a separate consent document. You do not need to consent to these additional studies in order to take part in this study.

### Other Information

### **COVID-19 Information**

To keep you, the study doctor, and the staff safe during the COVID-19 pandemic, some of your visits may be done by telephone or video conference, if available. Some of your tests or procedures may be done at a different visit or skipped. The study doctor will discuss these options with you, as needed. Tell your study doctor if you have any questions about visit requirements or options during the COVID-19 pandemic.

Some medications and treatments are not allowed while you are taking part in this study. It is very important that you tell the study doctor/study staff about all medicines (over-the-counter or prescription), herbal remedies, and supplements/vitamins you are taking or planning to take.

If you are taking medicines that affect your heart or change your stomach acid (like heartburn or indigestion medicine), you may need to stop taking these medicines. This will be discussed with you.

You cannot receive any other treatment for cancer while in this study. If you need surgery or radiation to help manage your care, this may be allowed if the doctor thinks it is safe to do so

You cannot receive a live vaccine while in this study. Some COVID-19 vaccines (such as the Moderna and Pfizer-BioNTech vaccines) are allowed. If you need a vaccine during the study, talk to the study doctor first.

#### 2. POSSIBLE RISKS

While on this study, you are at risk for side effects. These side effects will vary from person to person. The more commonly occurring side effects are listed in this form, as are rare but serious side effects. You should discuss these with the study doctor. You may also want to ask about uncommon side effects that have been observed in small numbers of patients but are not listed in this form. Many side effects go away shortly after treatment is stopped, but in some cases side effects may be serious, long-lasting or permanent, and may even result in hospitalization and/or death.

Tell the study staff about any side effects you may have, even if you do not think they are related to the study drug/procedures.

Nivolumab and sitravatinib may each cause low blood cell counts (red blood cells, platelets, and/or white blood cells):

- A low red blood cell count (anemia) may cause difficulty breathing and/or fatigue. You may need a blood transfusion.
- A low platelet count increases your risk of bleeding (such as nosebleeds, bruising, stroke, and/or digestive system bleeding). You may need a platelet transfusion.
- A low white blood cell count increases your risk of infection (such as pneumonia and/or severe blood infection). Infections may occur anywhere and become life-threatening. Symptoms of infection may include fever, pain, redness, and difficulty breathing.

# Sitravatinib Side Effects

# Common (occurring in 10% or more of patients)

- high blood pressurefatiguehand-foot syndrome(palms of hands/soles)
- nand-root syndrome (palms of hands/soles of feet having pain, swelling, and blistering)
- underactive thyroid gland (possible weight gain, heart failure, and/or constipation
- diarrhea
- nausea/vomiting
- inflamed and sore mouth
- loss of appetite
- weight loss

- abnormal liver tests (possible liver damage)
- abnormal amount of protein in the urine (possible kidney damage)
- hoarse voice

# Occasional (occurring in at least 5% but less than 10% of patients)

- dizziness
- skin rash
- abnormal blood test (possible pancreas damage/inflammation)
- abnormal salts, minerals, and/or acids in the blood (possible weakness, swelling, fatigue, low blood pressure, organ failure, heart problems, changes in mental status, and/or seizure)
- constipation
- change in taste
- abdominal pain
- dry mouth
- low blood cell counts (red, platelets)
- abnormal liver tests (possible liver damage

# Rare but serious (occurring in fewer than 5% of patients)

- stopping of the heart
- heart attack
- decreased brain function due to liver damage
- decrease in the pumping of the heart
- stroke
- · very high blood pressure
- blood clots, including those involving the lung
- abnormal EKG
- fatigue

- brain injury (possible headache, confusion, seizures, and/or vision loss)
- inflammation of the pancreas (possible abdominal pain)
- diarrhea
- weight loss
- nausea
- vomiting
- · decreased in appetite
- life-threatening stomach ulcer with tears in the stomach

- intestinal ulcer
- life-threatening bleeding
- kidney injury (possible fatigue, loss of appetite, confusion, nausea, and vomiting)
- inflammation of the colon or skin and inflammation of the colon, skin, thyroid, or heart muscle
- life-threatening infection

Drugs that are similar to sitravatinib also have been seen to cause difficulty healing wounds.

### Nivolumab Side Effects

# Common (occurring in more than 10%)

| fatigue/lack of energy | diarrhea | skin rash |
|------------------------|---------------------------|-----------|
| | <ul><li>itching</li></ul> | |

# Occasional (occurring in 3-10%)

- fever
- headache
- underactive thyroid gland (possible increased thyroid
- abnormal digestive blood test (possible inflammation of the pancreas)
- nausea/vomiting
- abnormal liver test
   (possible liver
   damage and/or
   yellowing of the eyes
   and/or skin)

- stimulating hormone lab test result, weight gain, heart failure, and/or constipation)
- overactive thyroid gland (possible decreased thyroid stimulating hormone lab test result, weight loss, heart rate changes, and/or sweating)
- abdominal pain
- loss of appetite
- low red blood cell count
- pain (including muscle/bone)
- lung inflammation (pneumonitis), and/or bronchitis (possible difficulty breathing)

# Rare (occurring in fewer than 3% of patients)

- fast heartbeat
- abnormal EKG
- heart inflammation/ inflammation of the tissue around the heart (possible chest pain)
- high blood pressure
- low blood pressure (possible dizziness and/or fainting)
- swelling of the brain (possible headache and/or mental status changes)
- inflammation of the brain and spinal cord (possible altered consciousness)
- inflammation of the membrane around the spinal cord and brain (possible headache and/or coma)
- swelling (face/arms/legs)
- chills
- difficulty sleeping
- dizziness
- dry/red skin
- hives
- skin blisters

- low blood levels of sodium (possible headache, confusion, seizures, and/or coma)
- abnormal blood test (possible pancreas damage)
- high blood sugar (possible diabetes)
- abnormal blood acid/base balance due to uncontrolled diabetes (possible organ damage)
- mouth blisters/sores (possible difficulty swallowing)
- constipation
- dehydration
- drv mouth
- inflammation of the intestines
- hole in the intestines or stomach (possibly leaking contents into the abdomen)
- liver inflammation
- liver failure/damage
- low blood cell count (platelets, white)
- viral/bacterial infection that affects nose,

- nerve damage (affecting the head and neck)
- muscle inflammation
- joint pain/stiffness
- dry eye
- blurry/double vision
- lung infiltrates (possible infection or inflammation)
- difficulty breathing (which can lead to respiratory failure)
- cough
- infusion reaction (possible fever, rash, pain, and/or swelling)
- immune response causing the body to attack itself (possibly causing muscle weakness)
- neuromuscular disease (possible weakness of eye, face, breathing and swallowing muscles) (myasthenic syndrome, myasthenia gravis)
- immune system reaction (possible fever, jaundice,

- very severe blistering skin disease (loss of large portion of skin and/or ulcers of the skin and digestive tract)
- red, dry, scaly patches of thickened skin (psoriasis)
- allergic skin reaction
- hair loss (partial or total)
- decreased production of adrenal hormones (possible weakness and/or low blood pressure)
- inflammation of the thyroid gland (possible tenderness in the neck)
- pituitary gland failure (possible hormone imbalance)
- blood vessel inflammation

- throat and airways (upper respiratory tract infection)
- destruction of red blood cells due to the body attacking itself (called autoimmune hemolytic anemia)
- abnormal kidney test (possible kidney damage)
- kidney failure
- breakdown of muscle tissue (possible kidney failure)
- Guillain-Barre syndrome--damage to the nervous system (causing numbness and/or paralysis)
- nerve damage (possible numbness, pain, and/or loss of motor function and/or "pins and needles" sensation)

- liver/spleen enlargement, irritability, and/or seizures)
- multi-organ disease causing lesions, most often in the lungs (sarcoidosis)
- allergic reaction, possibly lifethreatening (such as difficulty breathing, low blood pressure, and/or organ failure)
- flu-like symptoms
- patches of skin color loss
- inflammation of multiple areas of the body (see below)
- Hemophagocytic lymphohistiocytosis (HLH) syndrome (see below)

You may need to take drugs to reduce inflammation while taking nivolumab. Long-term use of these drugs may increase your risk of infection. These infections may occur anywhere and may be fatal. Treatment with antibiotic or antifungal drugs may be required to treat these infections.

At this time, it is not known whether taking a COVID-19 vaccine may affect the way that the study drug works in your body or if the study drug may affect the way the vaccine works in your body. No information is known about the interaction between a COVID-19 vaccine and nivolumab.

The study drug works by boosting the immune system. This may cause unknown side effects resulting from your immune system attacking your organs. This may cause inflammation and inflammation-related side effects in any organ or tissue.

Nivolumab may cause serious side effects that affect your immune system. Some of these side effects start as inflammation in different areas of the body like the skin, hormone glands, pancreas, pituitary gland, eye, kidney, or stomach. Tell the study staff right away if you have diarrhea, nausea, vomiting, blurred vision, dizziness, fainting, or you are feeling cold all the time.

Nivolumab may rarely cause Hemophagocytic lymphohistiocytosis (HLH) syndrome. HLH is a disease that may affect your body's defense system, (your immune system) and certain white blood cells made by your immune system may attack other blood

cells. These abnormal blood cells collect in your spleen and liver, causing these organs to enlarge, possibly causing fever, rash, and low blood cell counts.

### Frequency Unknown

- graft-versus-host disease (when transplanted donor tissue attacks the tissues of the recipient's body)
- Vogt Koyanagi Harada syndrome -- pigmented tissue (possible eye pain/swelling, hearing loss, and/or loss of skin color)
- risk of organ transplant rejection

**Using the study drugs together** may cause side effects that are not seen when each is given alone. The study drug combination may also increase the frequency and/or severity of the side effects listed above.

### **Other Risks**

**Blood draws** may cause pain, bleeding, and/or bruising. You may faint and/or develop an infection with redness and irritation of the vein at the site where blood is drawn. Frequent blood collection may cause anemia (low red blood cell count), which may create a need for blood transfusions.

**Questionnaires** may contain questions that are sensitive in nature. You may refuse to answer any question that makes you feel uncomfortable. If you have concerns about completing the questionnaire, you are encouraged to contact your doctor or the study chair.

**Fasting** may cause your blood sugar to drop. You may feel tired, hungry, and/or nauseous. If you have diabetes, it is important to talk to your doctor about managing your blood sugar while fasting.

**EKGs/ECHOs** may cause discomfort while lying on the exam table, and the tape on the EKG pads may cause skin irritation.

During the **MRI**, you may feel mild vibrations throughout your body. The machine will produce a loud knocking noise. This is normal. You will be given earplugs to protect your ears. Some people, especially those who tend to feel uncomfortable in small or closed spaces, may feel "closed in" and become anxious while in the scanner. The scanner has an intercom, which will allow you to speak to the staff during the procedure. If you feel ill or anxious during scanning, tell the MRI staff and the scanning will be stopped if you wish. The MRI will require a catheter to be inserted into one of your veins in order to inject the MRI contrast agent. This may cause skin irritation, bleeding, and/or infection. You may have an allergic reaction to the contrast agent.

The magnetic field used in MRI scanning may harm you if you have certain types of metal in your body (as might be found in pacemakers, neurostimulators, or certain clips). It may cause problems with devices, such as pacemakers. If you have metal in

your body or devices such as a pacemaker, you should discuss this with the study doctor.

Although every effort will be made to keep study data safe, there is a chance that your personal health information could be lost or stolen, which may result in a **loss of confidentiality**. You will read more about the protection of your information later in this form. Please ask the study doctor or study staff if you would like to know more about how your information will be protected while you are in this study.

A standard **bone scan** exposes you only to the radiation that comes from injecting the standard radioactive imaging solution for bone imaging.

CT scans send x-rays through the body at many different angles. You will be exposed to a small dose of radiation. All radiation adds up over a lifetime and may increase the risk of new cancer forming. Some people may feel "closed in" while lying in the scanner. However, the scanner is open at both ends, and an intercom allows you to talk with doctors and staff. If you feel ill or anxious during scanning, doctors and/or radiology technicians will give comfort, or the scanning will be stopped. Solution may also be given by vein to make the x-ray pictures more accurate. This may cause an uncomfortable feeling of warmth, nausea, and/or severe allergic reactions. The solution injection may also cause pain, bleeding, bruising, hives, and/or itching.

This study may involve unpredictable risks to the participants.

# **Pregnancy Related Risks**

Taking part in this study can result in risks to an unborn or breastfeeding baby, so you should not become pregnant, breastfeed a baby, or father a child while on this study. You must use birth control during the study if you are sexually active.

Birth Control Specifications: If you can become pregnant or father a child, you must use appropriate birth control methods, including a double-barrier method (2 methods at the same time), while you are on study and for 23 weeks (females) or 31 weeks (males) after you stop receiving the study drugs.

Your study doctor will discuss appropriate birth control methods with you.

Males: Tell the doctor right away if your partner becomes pregnant or suspects pregnancy.

Females: If you are pregnant, you will not be enrolled on this study. If you become pregnant or suspect that you are pregnant, you must tell your doctor right away.

Getting pregnant will result in your removal from this study.

### OPTIONAL PROCEDURES FOR THE STUDY

**Optional Procedure #1:** If you agree and the doctor thinks it is safe, you will have a tumor biopsy collected for biomarker testing, including genetic biomarkers, at screening, after 4 weeks of taking sitravatinib plus nivolumab, and at the end-of-

treatment on the study. The study doctor will tell you what kind of biopsy you will have. Biomarkers are found in the blood/tissue and may be related to your reaction to the study drug.

**Optional Procedure #2:** If you agree, blood (up to 10 tablespoons each time) will be drawn for biomarker testing, including genetic biomarkers, and other research tests that may help researchers understand the disease and/or your response to the study drugs (such as immune system and types of genetic testing). Blood will be drawn at screening, Week 4, Week 8, and at the end-of-treatment visit. You will not receive the results of these research tests.

You do not have to agree to the optional procedures in order to take part in this study. There are no benefits to you for taking part in the optional procedures. Future patients may benefit from what is learned. You may stop taking part at any time. There will be no cost to you for taking part in the optional procedures.

### **Optional Procedure Risks:**

Having **biopsies** performed may cause pain, bruising, bleeding, redness, low blood pressure, swelling, and/or infection at the site of the biopsies. An allergic reaction to the anesthetic may occur. A scar may form at the biopsy site. Rarely (in fewer than 3% of patients), major bleeding may occur.

**Blood draws** may cause pain, bleeding, and/or bruising. You may faint and/or develop an infection with redness and irritation of the vein at the site where blood is drawn. Frequent blood collection may cause anemia (low red blood cell count), which may create a need for blood transfusions.

### CONSENT/PERMISSION/AUTHORIZATION FOR OPTIONAL PROCEDURES

Circle your choice of "yes" or "no" for each of the following optional procedures:

Optional Procedure #1: Do you agree to have up to 3 biopsies for biomarker testing?

YES NO

**Optional Procedure #2:** Do you agree to have blood drawn up to 4 times for biomarker testing and research testing?

YES NO

### 3. COSTS AND COMPENSATION

If you suffer injury as a direct result of taking part in this study, MD Anderson health providers will provide medical care. However, this medical care will be billed to your insurance provider or you in the ordinary manner. You will not be reimbursed for expenses or compensated financially by MD Anderson or Mirati Therapeutics for this injury. You may also contact the Chair of MD Anderson's IRB at 713-792-6477 with questions about study-related injuries. By signing this consent form, you are not giving up any of your legal rights.

Certain tests, procedures, and/or drugs that you may receive as part of this study may be without cost to you because they are for research purposes only. However, your insurance provider and/or you may be financially responsible for the cost of care and treatment of any complications resulting from the research tests, procedures, and/or drugs. Standard medical care that you receive under this research study will be billed to your insurance provider and/or you in the ordinary manner. Before taking part in this study, you may ask about which parts of the research-related care may be provided without charge, which costs your insurance provider may pay for, and which costs may be your responsibility. You may ask that a financial counselor be made available to you to talk about the costs of this study.

Samples that are collected from you in this study may be used for the development of treatments, devices, new drugs, or patentable procedures that may result in commercial profit.

There are no plans to compensate you for any patents or discoveries that may result from your participation in this research.

You will receive no compensation for taking part in this study.

### **Additional Information**

- 4. You may ask the study chair (Dr. Pavlos Msaouel, at 713-563-4585) any questions you have about this study. You may also contact the Chair of MD Anderson's Institutional Review Board (IRB a committee that reviews research studies) at 713-792-6477 with any questions that have to do with this study or your rights as a study participant.
- 5. You may choose not to take part in this study without any penalty or loss of benefits to which you are otherwise entitled. You may also withdraw from participation in this study at any time without any penalty or loss of benefits. If you decide you want to stop taking part in the study, it is recommended for your safety that you first talk to your doctor who can then decide if you need to have any visits or tests to check on your health.. If you withdraw from this study, you can still choose to be treated at MD Anderson.

If you stop being in the research, already collected data may not be removed from the study database. You may be asked whether the study doctor can collect data from your routine medical care. If you agree, this data will be handled the same as research data.

- 6. This study or your participation in it may be changed or stopped without your consent at any time by the study chair, Mirati Therapeutics, BMS, the U.S. Food and Drug Administration (FDA), the Office for Human Research Protections (OHRP), or the IRB of MD Anderson.
- 7. You will be informed of any new findings or information that might affect your willingness to continue taking part in the study, including the results of all of your standard tests performed as part of this research, and you may be asked to sign another informed consent and authorization form stating your continued willingness to participate in this study.

The results for most of the tests required in this study will be placed in your medical record. However, you will not receive the results of research (correlative) studies.

- 8. MD Anderson may benefit from your participation and/or what is learned in this study.
- This study is sponsored and/or supported by: Mirati Therapeutics and Bristol Myers-Squibb (BMS).
- 10. In a medical emergency, you may be cared for by someone who has a financial interest with the study sponsor(s)/supporter. If you have any questions about this, you may call the IRB at 713-792-6477.

### **Future Research**

### Data

Your personal information is being collected as part of this study. These data may be used by researchers at MD Anderson, Mirati Therapeutics, BMS, and/or shared with other researchers and/or institutions for use in future research.

#### Samples

Samples (such as blood and/or tissue) are being collected from you as part of this study. Researchers at MD Anderson may use any leftover samples that are stored at MD Anderson in future research.

Before being used or shared for future research, every effort will be made to remove your identifying information from any data and/or research samples. If all identifying information is removed, you will not be asked for additional permission before future research is performed.

In some cases, all of your identifying information may not be removed before your data or research samples are used for future research. If future research is performed at MD Anderson, the researchers must get approval from the Institutional Review Board (IRB) of MD Anderson before your data and/or research samples can be used. At that time, the IRB will decide whether or not further permission from you is required. The IRB is a committee of doctors, researchers,

and community members that is responsible for protecting study participants and making sure all research is safe and ethical.

If this research is not performed at MD Anderson, MD Anderson will not have oversight of any data and/or samples.

If you do not want your samples or data to be used for future research, tell the study doctor. You may withdraw your samples at any time by telling your study team. If you decide to withdraw your samples, they will be returned to the lab they came from or destroyed. However, the data and test results already collected from your samples will be kept and may be used.

### **Genetic Research**

Research samples collected from you as part of this study may be used for genetic research, which may include whole genome sequencing. Whole genome sequencing is a type of testing in which researchers study your entire genetic makeup (DNA). This may help researchers learn how changes in the ordering of genes may affect a disease or response to treatment. If genetic research is done with your samples, those who have access to those samples may be able to identify you. The results of this research may also be able to be linked to you. The same level of data protection that covers your individual data does not apply to summary results (when data from the whole study is combined).

A federal law, called the Genetic Information Nondiscrimination Act (GINA), generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. This law generally will protect you in the following ways:

- Health insurance companies and group health plans may not request your genetic information that we get from this research.
- Health insurance companies and group health plans may not use your genetic information when making decisions regarding your eligibility or premiums.
- Employers with 15 or more employees may not use your genetic information that we get from this research when deciding to hire, promote, or fire you or when setting the terms of your employment.

Be aware that this federal law does not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. Nor does this federal law prohibit discrimination based on an already known genetic disease or disorder.

### **Outside Care**

Part of your care may be provided outside of MD Anderson by your home doctor(s).

# **Conflict of Interest**

Dr. Pavlos Msaouel (Study Chair) has received compensation from BMS as a Consultant. The financial interests are within the limits of the conflict of interest policy.

Dr. Nizar Tannir (Co-Investigator) has received compensation from BMS as a Consultant. The financial interests are within the limits of the conflict of interest policy.

### <u>Authorization for Use and Disclosure of Protected Health Information (PHI):</u>

- A. During the course of this study, MD Anderson will be collecting and using your PHI, including identifying information, information from your medical record, and study results. For legal, ethical, research, and safety-related reasons, your doctor and the research team may share your PHI with:
  - Federal agencies that require reporting of clinical study data (such as the FDA, National Cancer Institute [NCI], and OHRP)
  - The IRB and officials of MD Anderson
  - Mirati Therapeutics, who is the supporter of this study, along with Bristol-Myers Squibb, and/or any future sponsors/supporters of the study
  - Study monitors and auditors who verify the accuracy of the information
  - Individuals who put all the study information together in report form
  - Other participating study sites

Study sponsors and/or supporters receive limited amounts of PHI. They may also view additional PHI in study records during the monitoring process. MD Anderson's contracts require sponsors/supporters to protect this information and limit how they may use it.

The results of this research may be published in scientific journals or presented at medical meetings, but your identity will not be disclosed.

- B. Signing this consent and authorization form is optional but you cannot take part in this study or receive study-related treatment if you do not agree and sign.
- C. MD Anderson will keep your PHI confidential when possible (according to state and federal law). However, in some situations, the FDA could be required to reveal the names of participants.
  - Once disclosed outside of MD Anderson, federal privacy laws may no longer protect your PHI.
- D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected.

| E. | A description of this clinical trial will be available on http://www.ClinicalTrials.gov, |
|---|---|
| | as required by U.S. Law. This Web site will not include information that can identify |
| | you. At most, the Web site will include a summary of the results. You can search |
| | this Web site at any time |

# **CONSENT/AUTHORIZATION**

I understand the information in this consent form. I have had a chance to read the consent form for this study, or have had it read to me. I have had a chance to think about it, ask questions, and talk about it with others as needed. I give the study chair

| permission to enroll me on this study. By signing this consent form, I any of my legal rights. I will be given a signed copy of this consent do | |
|---|---|
| SIGNATURE OF PARTICIPANT | DATE |
| PRINTED NAME OF PARTICIPANT | |
| LEGALLY AUTHORIZED REPRESENTATIVE (LAR) The following signature line should only be filled out when the partic the capacity to legally consent to take part in the study and/or sign the or her own behalf. | • |
| SIGNATURE OF LAR | DATE |
| PRINTED NAME and RELATIONSHIP TO PARTICIPANT | |
| WITNESS TO CONSENT I was present during the explanation of the research to be performed 2021-0057. | under Protocol |
| SIGNATURE OF WITNESS TO THE VERBAL CONSENT PRESENTATION (OTHER THAN PHYSICIAN OR STUDY CHAIR) A witness signature is only required for non-English speakers utilizing the short form consent process (VTPS) and patients who are illiterate. | DATE |
| PRINTED NAME OF WITNESS TO THE VERBAL CONSENT | |
| PERSON OBTAINING CONSENT I have discussed this research study with the participant and/or his or representative, using language that is understandable and appropriat have fully informed this participant of the nature of this study and its pand risks and that the participant understood this explanation. | e. I believe that I |
| PERSON OBTAINING CONSENT | DATE |
| PRINTED NAME OF PERSON OBTAINING CONSENT | |

Protocol 2021-0057 November 30, 2022 Page 17 of 17

| TRANSLA' | <b>TOR</b> |
|----------|------------|
|----------|------------|

| I have translated the above | informed consent as written (without add | ditions or |
|---|---|---|
| subtractions) into | and assisted | and assisted the people |
| , <u>(</u> 1 | Name of Language) | |
| obtaining and providing conscious consent process for this part | sent by translating all questions and resp<br>ticipant. | onses during the |
| NAME OF TRANSLATOR | SIGNATURE OF TRANSLATOR | DATE |
| | translator was a member of the research<br>nslator, must sign the witness line.) | n team. (If checked, |